CLINICAL TRIAL: NCT06677073
Title: Effects of Maximal Fat Oxidation Exercise and High-intensity Interval Training on Fat Loss in Overweight Young Women
Brief Title: Effects of FATmax Exercise and HIIT on Fat Loss in Overweight Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EOMFOEAHITOFLIOYW
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Overweight
Keywords: High-intensity interval training; Maximal fat oxidation; Overweight; Fat loss; Female
MeSH Terms: conditions — Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIIT group (Experimental)
  Interventions: Behavioral: High-intensity interval training
- FATmax group (Experimental)
  Interventions: Behavioral: Maximal fat oxidation exercise

INTERVENTIONS:
Behavioral: High-intensity interval training — High-intensity interval training
  Arms: HIIT group
Behavioral: Maximal fat oxidation exercise — Maximal fat oxidation exercise
  Arms: FATmax group

SUMMARY:
This study investigated the effects of two exercise modalities: high-intensity interval training (HIIT) and maximal fat oxidation (FATmax) exercise on fat loss in overweight young women. Participants were randomly assigned to either the HIIT or FATmax group, underwent an 8-week supervised exercise intervention.

DETAILED DESCRIPTION:
This study aims to compare the effects of HIIT and FATmax exercise on fat loss in overweight young women. Participants were recruited and randomly assigned to either the HIIT group or the FATmax group. The intervention lasted for 8 weeks, during which participants maintained their usual diet. Both body morphology and body composition were assessed before and after the intervention. In order to recommend exercise strategy for overweight young women reduce fat and improve their health.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged between 18 and 30 years.
* Overweight, BMI greater than 24.0 kg·m-2.
* Participants Lack of exercise habits.
* Participants Without significant fluctuation in weight.

Exclusion Criteria:

* Participants took drugs affecting metabolism and hormones during the experimental period.
* Participants had a history of oral weight loss pills and contraceptive pills.
* Participants had a history of smoking, alcohol consumption, or daily consumption of caffeine-containing beverages.
* Participants had cardiovascular or basal metabolic disorders, such as hypertension, coronary heart disease, or diabetes mellitus.
* Participants had other acute or chronic injuries related to exercise.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 8 weeks
  The change of body weight before and after intervention.
Body mass index (BMI) | 8 weeks
  The change of body mass index before and after intervention.
Waist circumference | 8 weeks
  The change of waist circumference before and after intervention.
Hip circumference | 8 weeks
  The change of hip circumference before and after intervention.
Body fat weight | 8 weeks
  The change of body fat weight before and after intervention.
Body fat percentage | 8 weeks
  The change of body fat percentage before and after intervention.
Visceral fat area | 8 weeks
  The change of visceral fat area before and after intervention.

SECONDARY OUTCOMES:
Height | 8 weeks
  The change of height before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No